CLINICAL TRIAL: NCT00358878
Title: Satavaptan Cirrhotic Ascites Treatment Study: a Double-blind, Randomised, Parallel-group Comparison of Treatment With Satavaptan at 5 to 10 mg Daily Versus Placebo on Top of Conventional Treatment in Patients With Ascites Due to Cirrhosis of the Liver
Brief Title: Cirrhotic Ascites Treatment With Satavaptan in Patients With Ascites Due to Cirrhosis of the Liver (CATS)
Acronym: CATS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4492; EudraCT : 2006-000132-27; LTS10036
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Ascites; Liver Cirrhosis
Keywords: Ascites; Liver Cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Satavaptan (Experimental)
  Interventions: Drug: Satavaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Satavaptan — oral administration once daily
  Other Names: SR121463B
  Arms: Satavaptan
Drug: placebo — oral administration once daily
  Arms: Placebo

SUMMARY:
Primary:To evaluate the efficacy of satavaptan on top of conventional treatment in the treatment of clinically evident ascites in participants with cirrhosis of the liver.

Secondary:To evaluate the tolerability and safety of satavaptan over a 52-week treatment period in participants with cirrhosis of the liver and ascites.

The one-year double blind placebo controlled period is extended up to 2 years in a long term safety study (PASCCAL-2).

ELIGIBILITY:
Inclusion Criteria:

* Participants with cirrhosis of the liver
* Participants with clinically evident ascites primarily managed by diet and/or diuretics
* Stable treatment of ascites for at least the previous 2 weeks without paracentesis
* Participants having undergone no more than one therapeutic paracentesis in the previous 6 months.

Exclusion Criteria:

* Participants with an existing functional transjugular intrahepatic portosystemic shunt (TIPS) or other shunt
* Known hepatocellular carcinoma
* Participants with ascites of cardiac origin or due to peritoneal infection (e.g. tuberculosis) or peritoneal carcinoma
* Participants previously exposed to satavaptan in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of ascites worsening | at week 12

SECONDARY OUTCOMES:
Composite endpoint of ascites worsening | at week 24
Increase in ascites | at week 12

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (21):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Madrid, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Wong F, Watson H, Gerbes A, Vilstrup H, Badalamenti S, Bernardi M, Gines P; Satavaptan Investigators Group. Satavaptan for the management of ascites in cirrhosis: efficacy and safety across the spectrum of ascites severity. Gut. 2012 Jan;61(1):108-16. doi: 10.1136/gutjnl-2011-300157. Epub 2011 Aug 11. PMID 21836029